CLINICAL TRIAL: NCT01701999
Title: Phase 2b, Two-part, Open-label, Uncontrolled Study to Evaluate Safety, Tolerability, and Immunogenicity of a Single 40-µg Dose of Recombinant Botulinum Vaccine A/B (rBV A/B) for the Production of BabyBIG® in Volunteers Previously Immunized With Pentavalent Botulinum Toxoid for Occupational Protection
Brief Title: Safety, Tolerability, and Immunogenicity Study of Investigational Recombinant Botulinum Vaccine A/B (rBV A/B) in Volunteers Previously Immunized With Investigational Pentavalent Botulinum Toxoid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: California Department of Public Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: rBV A/B-CL-001
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Results first posted 2017-02-09 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Botulism
Keywords: Botulism Vaccine
MeSH Terms: conditions — Botulism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine (Experimental)
  Interventions: Biological: rBV A/B

INTERVENTIONS:
Biological: rBV A/B — rBV A/B injections will consist of a single 40 µg injection of total antigen (20 µg of Antigen A and 20 µg of Antigen B) adsorbed to 0.2% (wt/vol) Alhydrogel™, in a total dose volume of 0.5 mL. The vaccine will be administered by intramuscular injection in the deltoid muscle, preferably in the nondominant arm.

SUMMARY:
Study rBV A/B-CL-001 is a Phase 2b, 2-part, open-label, uncontrolled study to evaluate safety, tolerability, and immunogenicity of a single dose of recombinant botulinum vaccine A/B (rBV A/B) for the production of BabyBIG in volunteers previously immunized with the pentavalent botulinum (PBT) toxoid. This study is designed to determine neutralizing antibody levels for botulinum toxin types A and B in healthy subjects who were previously immunized with the PBT for occupational protection and who receive the rBV A/B. Subjects with titers of the neutralizing antibodies against the toxins would be candidates for plasma donation for BabyBIG production.

ELIGIBILITY:
Inclusion Criteria:

* The volunteer has received pentavalent botulinum toxoid for occupational protection under BB IND 0161, with the previous pentavalent botulinum toxoid dose at least 6 months prior to the planned rBV A/B dose.
* The volunteer is between the ages of 18 and 69 years at the time of consent.
* The volunteer is healthy and has an acceptable medical history.
* The volunteer meets the subject suitability requirements and recommendations for source plasma donors (for Part 2 subjects only).
* The volunteer, if female and of childbearing potential, is not pregnant or lactating, and agrees to use an acceptable form of FDA-approved contraception for the duration of the study.
* The volunteer has the ability to understand the requirements of the study and provide informed consent.
* The volunteer agrees to complete the subject diary on a daily basis for 7 days post-vaccination and to report concomitant medication and adverse events during the study period.
* The volunteer provides written authorization for use and disclosure of protected health information.
* The volunteer agrees not to donate blood or blood products (outside of study procedures) during the course of the study.
* The volunteer has personal health insurance.

Exclusion Criteria:

* Be pregnant or nursing
* The volunteer has a history of laboratory evidence of syphilis, acquired immunodeficiency syndrome, Creutzfeldt-Jakob disease, or infection with human immunodeficiency viruses 1 or 2, human T cell lymphotropic virus 1, hepatitis B virus, or hepatitis C virus.
* The volunteer had prior severe local or severe systemic reaction to last immunization with pentavalent botulinum toxoid.
* The volunteer has a known allergy to aluminum compounds, yeast, or other components of the vaccine.
* The volunteer has donated one or more units of blood or undergone plasmapheresis within 28 days before screening.
* The volunteer has received a blood product or immunoglobulin within 6 months of screening or plans to receive such products during the study.
* The volunteer has received licensed nonliving vaccine within 14 days before study entry or licensed live vaccine within 60 days before study entry.
* The volunteer has received investigational products (drugs, biologics, vaccines, or implantable devices) 60 days prior to study entry or plans to receive experimental products at any time during the study.
* The volunteer has received prescription immunosuppressive or immunomodulatory agents, including parenteral, inhaled, or oral corticosteroids within 3 months before screening or plans on receiving such therapy at any time during the study with the exceptions (Subjects who have used prescription topical steroids may be enrolled 2 weeks after the therapy is completed; Intra-articular, bursal, or tendon injectable steroids are permitted; Any over-the-counter topical steroid use is permitted; Ophthalmic and intranasal steroids are permitted).
* The volunteer has received cytotoxic therapy at any time in the previous 5 years to study entry.
* The volunteer has an active systemic or recurrent disease that would place the subject at unacceptable risk of injury, require hospitalization, or require surgical intervention.
* The volunteer has a history of alcohol or drug abuse within 12 months before screening.
* The volunteer has past, present, or suspected illicit injection drug use.
* The volunteer has inflammatory, vasculitic, or rheumatic disease, including systemic lupus erythematosus, polymyalgia rheumatica, rheumatoid arthritis, or scleroderma.
* The volunteer has clinically recognized hepatic or renal insufficiency.
* The volunteer has uncontrolled hypertension.
* The volunteer has moderate to severe asthma, chronic obstructive pulmonary disease, or other significant pulmonary disease.
* The volunteer has a seizure disorder.
* The volunteer has moderate or severe illness or oral temperature of 100.4°F or greater within 3 days prior to immunization.
* The volunteer is determined by the investigator to be unsuitable for participation in this trial for any reason.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen S. Arnon, M.D., Principal Investigator — California Department of Public Health
Locations (2):
- United States (2):
  - California Department of Public Health, Richmond, California
  - Battelle Biomedical Research Center, West Jefferson, Ohio

REFERENCES:
- [Derived] Khouri JM, Motter RN, Arnon SS. Safety and immunogenicity of investigational recombinant botulinum vaccine, rBV A/B, in volunteers with pre-existing botulinum toxoid immunity. Vaccine. 2018 Apr 5;36(15):2041-2048. doi: 10.1016/j.vaccine.2018.02.042. Epub 2018 Feb 21. PMID 29475762
- See also: Related Info — http://www.infantbotulism.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Initial Safety and Immunogenicity (Part 1): Part 1 included scheduled assessments of the safety and immunogenicity of a single 40 µg dose of rBV A/B over a 12-week period with a safety follow-up at 6 months.
- Safety, Immunogenicity, and Plasma Collection (Part 2): Part 2 was conducted to collect source plasma for potential use in the production of BabyBIG® and to assess safety and immunogenicity of a single 40 µg dose of over a 12-week period; Part 2 included a follow-up for safety assessment at 6 months. Participants in Part 2 did not participate in Part 1.
Period: Overall Study
Arm/Group | Initial Safety and Immunogenicity (Part 1) | Safety, Immunogenicity, and Plasma Collection (Part 2)
Started | 8 | 37
Completed | 8 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Initial Safety and Immunogenicity (Part 1) | Safety, Immunogenicity, and Plasma Collection (Part 2) | Total
Number analyzed (Participants) | 8 | 37 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (13.5) | 44.0 (10.7) | 45.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 20 | 23
  Male | 5 | 17 | 22

OUTCOME MEASURES:

1. Primary Outcome: Four-Fold Increase in Neutralizing Antibody Concentration (NAC)
Description: Proportion of participants achieving a four-fold or greater increase in NAC up to Week 4 compared with Week 0 for both botulinum toxin A and toxin B (a proportion ≥ 0.50 was considered a success).
Time Frame: Week 0 to Week 4
Measure: Number; unit: proportion of participants
Arm/Group | Initial Safety and Immunogenicity (Part 1) | Safety, Immunogenicity, and Plasma Collection (Part 2)
Number analyzed (Participants) | 8 | 37
proportion of participants
  Type A | 0.75 | 0.84
  Type B | 0.75 | 0.89

2. Secondary Outcome: Three-Fold Increase in Neutralizing Antibody Concentration (NAC)
Description: Proportion of participants achieving a three-fold or greater increase in NAC up to Week 4 compared with Week 0 for both botulinum toxin A and toxin B (a proportion ≥ 0.50 was considered a success)
Time Frame: Week 0 to Week 4
Measure: Number; unit: proportion of participants
Arm/Group | Initial Safety and Immunogenicity (Part 1) | Safety, Immunogenicity, and Plasma Collection (Part 2)
Number analyzed (Participants) | 8 | 37
proportion of participants
  Type A | 0.75 | 0.95
  Type B | 0.75 | 0.89

3. Secondary Outcome: Two-Fold Increase in the Area Under the Neutralizing Antibody Concentration (NAC) Curve
Description: Proportion of participants achieving a two-fold increase in the area under the plasma NAC-time curve between Week 0 and Week 12 in comparison with a straight-line extension of the Week 0 NAC to Week 12 for both botulinum toxin A and toxin B. A proportion ≥ 0.50 was considered a success.
Time Frame: Week 0 to Week 12
Measure: Number; unit: proportion of participants
Arm/Group | Initial Safety and Immunogenicity (Part 1) | Safety, Immunogenicity, and Plasma Collection (Part 2)
Number analyzed (Participants) | 8 | 37
proportion of participants
  Type A | 0.75 | 0.95
  Type B | 0.88 | 0.89

4. Other Pre Specified Outcome: Collected Plasma Volume
Description: Measurement of the volume of source plasma containing neutralizing antibodies against botulinum toxin type A and type B collected by plasmapheresis in Part 2.
Time Frame: Week 1 to Week 12
Population: Participants in Part 1 were only analyzed for safety data, and one participant in Part 2 was excluded from plasma collection due to not meeting the plasma donor minimum weight requirement.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Initial Safety and Immunogenicity (Part 1) | Safety, Immunogenicity, and Plasma Collection (Part 2)
Number analyzed (Participants) | 0 | 36
mL |  | 13463.3 (4440.5)

ADVERSE EVENTS:
Time Frame: Six months following rBV A/B administration
Description: Adverse events (AEs) indicated with * were largely classified as treatment-related reactions (TRRs). Of the 32 and 186 total AEs in Parts 1 and 2, respectively, 21 (65.6%) and 117 (62.9%) were TRRs within the indicated categories. Also, of the 21 and 117 TRRs in Parts 1 and 2, respectively, 19 (90.5%) and 97 (82.9%) occurred within 7 days of the rBV A/B injection, and 8 of 8 participants in Part 1 (100%) and 30 of 37 in Part 2 (81.1%) had at least one TRR within 7 days of the rBV A/B injection.
Arm/Group | Initial Safety and Immunogenicity (Part 1) | Safety, Immunogenicity, and Plasma Collection (Part 2)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/37
Other Adverse Events (participants affected / at risk) | 8/8 | 34/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Safety and Immunogenicity (Part 1) (N=8) | Safety, Immunogenicity, and Plasma Collection (Part 2) (N=37)
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Nausea* (Gastrointestinal disorders) | 0 | 3
Chills* (General disorders) | 0 | 2
Injection site anaesthesia* (General disorders) | 1 | 0
Injection site erythema* (General disorders) | 5 | 19
Injection site induration* (General disorders) | 0 | 3
Injection site nodule* (General disorders) | 0 | 2
Injection site pain* (General disorders) | 6 | 15
Injection site papule (General disorders) | 1 | 0
Injection site pruritus* (General disorders) | 3 | 9
Injection site reaction* (General disorders) | 1 | 0
Injection site swelling* (General disorders) | 3 | 18
Injection site urticaria* (General disorders) | 0 | 1
Malaise* (General disorders) | 0 | 5
Pain* (General disorders) | 0 | 1
Pyrexia* (General disorders) | 0 | 2
Swelling* (General disorders) | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Infusion site hematoma (Injury, poisoning and procedural complications) | 0 | 1
Injection site swelling* (Injury, poisoning and procedural complications) | 0 | 1
Procedural complication* (Injury, poisoning and procedural complications) | 0 | 14
Procedural pain (Injury, poisoning and procedural complications) | 0 | 3
Aspartate aminotransferase increased* (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 1 | 0
Body temperature increased* (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 5
Haemaglobin decreased (Investigations) | 1 | 1
Haemaglobin increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Protein total decreased (Investigations) | 0 | 2
Urine ketone body present (Investigations) | 0 | 1
Muscle spasms* (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness* (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain* (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia* (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Sensation of heaviness* (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache* (Nervous system disorders) | 0 | 5
Paraesthesia* (Nervous system disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema* (Skin and subcutaneous tissue disorders) | 0 | 4
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous* (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Sunburn (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria* (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes